CLINICAL TRIAL: NCT00191178
Title: Pilot Study Investigating the Effects of Insulin Lispro Low Mixture Therapy Compared With Insulin Glargine on Perceived Mood Symptoms in Patients With Type 2 Diabetes Mellitus
Brief Title: Effects of Insulin in Perceived Mood Symptoms in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 4957; F3Z-MC-IOOC
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-10-13 (Estimated); Status verified 2010-10

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Insulin Glargine

INTERVENTIONS:
Drug: insulin lispro protamine suspension:insulin lispro rDNA origin low mix
Drug: insulin glargine

SUMMARY:
This study investigates the influence of two different insulin regimens, twice-daily insulin lispro low mix (LM) and once-daily insulin glargine, on perceived physical, mood, and cognitive symptoms as well as cognitive-motor task performance in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed as having type 2 diabetes mellitus, as defined by the World Health Organization
* Are being treated with metformin therapy alone, metformin therapy plus once-daily insulin, or metformin plus one or more other oral antihyperglycemic agents at the time of study entry
* Female patients not breastfeeding and female patients of childbearing potential must test negative for pregnancy at time of study entry based on a urine pregnancy test and do not intend to become pregnant during the study and agree to use a reliable form of birth control during the study
* Hemoglobin A1c greater than or equal to 7.0% and less than or equal to 10% within 3 months prior to visit 1
* Have given informed consent to participate in the study in accordance with local regulations

Exclusion Criteria:

* Are investigator site personnel directly affiliated with the study, or are immediate family of investigator site personnel directly affiliated with the study.
* Have received treatment within the last 30 days with a drug that has not received regulatory approval for any indication at the time of study entry
* Have previously been diagnosed with clinical depression or have been treated with a central nervous system stimulant, antidepressant, antipsychotic, or anxiolytic agent within 30 days prior to study entry
* Have a known allergy to insulin lispro low mixture, insulin glargine, metformin hydrochloride, or excipients contained in these products
* Have known hypersensitivity or contraindication to metformin hydrochloride

Ages: 21 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2003-08; Study Completion 2005-07

PRIMARY OUTCOMES:
Compare twice-daily insulin lispro Low Mix therapy and once-daily insulin glargine therapy with respect to perceived mood on patient-rated questionnaires following chronic treatment administration in patients with type 2 diabetes
Instruments used/tests performed:hand held computers to rate a series of 13 symptoms;hand held computers to administer a series of cognitive-motor performance tests;blood glucose testing

SECONDARY OUTCOMES:
Compare insulin lispro Low Mix therapy and insulin glargine therapy with respect to:scores (collective and specific) on patient-rated mood, physical, and cognitive symptoms;scores on specific cognitive-motor performance tests
physical energy level as reflected by subjective symptoms, self-report of activity level, and physical motion as reflected by a pedometer worn at the waist
specific measures of depression, according to the Beck Depression Inventory-II
blood glucose rate of change;eight-point self-monitored blood glucose profile;episodes of hypoglycemia, including episodes of severe hypoglycemia

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Monday-Friday 9am-5pm Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST) or speak with your personal physician, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Cox DJ, McCall A, Kovatchev B, Sarwat S, Ilag LL, Tan MH. Effects of blood glucose rate of changes on perceived mood and cognitive symptoms in insulin-treated type 2 diabetes. Diabetes Care. 2007 Aug;30(8):2001-2. doi: 10.2337/dc06-2480. Epub 2007 May 1. No abstract available. PMID 17473060
- [Derived] Cox DJ, Ford D, Gonder-Frederick L, Clarke W, Mazze R, Weinger K, Ritterband L. Driving mishaps among individuals with type 1 diabetes: a prospective study. Diabetes Care. 2009 Dec;32(12):2177-80. doi: 10.2337/dc08-1510. PMID 19940224